CLINICAL TRIAL: NCT03799172
Title: Echinocandins Versus Azoles as First-line Therapy for the Treatment of Candidemia in Intensive Care Units
Brief Title: Echinocandins Versus Azoles for Candidemia Treatment
Acronym: AntiCandiTreat
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2019_001
Record Dates: First submitted 2019-01-03; First posted 2019-01-10 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Candidemia
MeSH Terms: conditions — Candidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Echinocandin group: Echinocandin group is the group of patients who received echinocandins as first-line therapy for candidemia
  Interventions: Drug: Echinocandin treatment
- Triazole group: Triazole group is the group of patients who received triazoles as first-line therapy for candidemia
  Interventions: Drug: Triazole treatment

INTERVENTIONS:
Drug: Echinocandin treatment — Patients received echinocandins as a first-line therapy after candidemia diagnosis according to the standard of care
  Groups: Echinocandin group
Drug: Triazole treatment — Patients received triazoles as a first-line therapy after candidemia diagnosis according to the standard of care.
  Candidemia was defined as at least one blood culture positive for Candida.
  Groups: Triazole group

SUMMARY:
Candidemia is the most frequent invasive fungal disease in intensive care units (ICUs). It remains a major health concern, considering its attributable mortality up to 40% in critically ill patients. Successful clinical outcome requires early diagnosis and effective antifungal therapy. Guidelines for the treatment of candidemia were published by the Infectious Diseases Society of America (IDSA) and the European Society of Clinical Microbiology and Infectious Diseases (ESCMID). According to these guidelines, echinocandins are the preferred first-line therapy for candidemia in critically ill patients. Considering the bibliography supporting this statement, the place of triazoles still needs to be defined in candidemia therapeutic arsenal. In this context, we are setting up a retrospective cohort study using Hospital database to compare the efficacy of echinocandins and azoles for the treatment of candidemia in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a diagnosis of candidemia during ICU stay and were treated with echinocandins or azoles

Exclusion Criteria:

* Patients with neutropenia
* Patients without antifungal treatment
* Patients who received antifungal therapy for more than two days before candidemia diagnosis
* Patients receiving liposomal amphotericin b or multiple antifungal agents as first-line therapy
* Patients who received less than 4 days of antifungal therapy after candidemia diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of candidemia during their ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of all cause hospital mortality on day 90 between echinocandins and azoles | Mortality on day 90 after antifungal initiation
  Comparison of all cause hospital mortality on day 90 between echinocandins and azoles

SECONDARY OUTCOMES:
Comparison of treatment success on day 30 between echinocandins and azoles. | Treatment success on day 30 after antifungal initiation
  Treatment success is defined as a complete response if the following two criteria were full-filled: survival and resolution of all attributable symptoms and signs of disease, and mycological success (documented clearance of pathogen from the blood).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Hôpital de la Croix-Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided